CLINICAL TRIAL: NCT00280787
Title: LCCC 0215: Induction Chemotherapy Using Paclitaxel, Carboplatin, CPT-11 With Pegfilgrastim Support Followed by Conformal Radiotherapy and Paclitaxel/Carboplatin/ZD1839 in Locally Advanced Unresectable Stage IIIA/B Non-Small Cell Carcinoma of the Lung
Brief Title: Induction Chemotherapy Using Paclitaxel, Carboplatin, CPT-11 With Pegfilgrastim
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0215; NCT00522366 (obsolete NCT alias)
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: unresectable; induction; radiotherapy; ZD1839
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Irinotecan; pegfilgrastim; Radiotherapy, Conformal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m2 administered on Day 1, of a 21 day cycle. Subjects will receive 2 cycles
  Other Names: Taxol
Drug: Carboplatin — Area Under the Curve(AUC)=5 administered on Day 1 of a 21 day cycle. Subjects will receive 2 cycles.
  Other Names: Paraplatin
Drug: CPT-11 — 100 mg/m2 administered on Day 1 of each 21 day cycle. Subjects will receive 2 cycles.
  Other Names: Irinotecan
Drug: Pegfilgrastim — 6 mg administered on Day 2 each each 21 day cylce. Subjects will receive 2 cycles of treatment.
  Other Names: Neulasta
Radiation: Conformal radiotherapy — Radiation therapy will be administered with standard daily fractionation of 2.0 Gy per fraction, 5 days per week.The total dose of radiotherapy will be 74 Gy

SUMMARY:
Patients enrolled on this study will have been diagnosed with non-small cell lung cancer which cannot be removed by an operation. The standard treatment for this disease is a combination of chemotherapy and radiation therapy; however, the best way to combine these treatments is not known. This study will examine if the combination of chemotherapy and radiotherapy has an increased effect on slowing tumor growth with the addition of a drug called ZD1839.

In this study, chemotherapy will be given initially (induction therapy) to try to control the spread of the cancer. Then radiation and chemotherapy will be given together. Receiving chemotherapy at the same time as radiation treatments can enhance the effect of the radiation. In this study, patients will receive a drug called ZD1839. In laboratory tests on cancer cells, ZD1839 has shown an additive effect when used in combination with radiation. ZD1839 has also been shown to slow or stop growth in tumors.

The purpose of this study is to determine the side effects and effectiveness of using ZD1839 when used with radiation in this treatment regimen (induction chemotherapy followed by combination chemotherapy, ZD1839, and radiation therapy).

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality in the United States. In 2002, approximately 170,000 new cases of lung cancer will be diagnosed, and approximately 160,000 deaths will occur. Eighty percent of cases of lung cancer are of the non-small cell type, and 30 to 35% will be Stage IIIA/B and are considered potentially curable. The standard of care in the United States for those patients with unresectable Stage IIIA/B and a good performance status (PS) is a combination of systemic chemotherapy and thoracic radiation therapy (TRT). What is not clear in the management of these patients is the optimal strategy to employ in the combined-modality approach, as well as the optimal chemotherapy and radiation therapy dose and schedule.

Induction and Concurrent Chemoradiation Therapy for Stage IIIA/B NSCLC The use of combined modality has become the standard of care in unresectable Stage IIIA/B non-small cell lung cancer (NSCLC). In the curative approach to this disease, both local control and eradication of occult micrometastatic disease must be achieved. Combined-modality trials employing induction chemotherapy have suggested a reduction in the rate of metastatic disease, suggesting that effectively delivered chemotherapy can eradicate occult micrometastatic disease. All of the trials cited have shown improved survival for the combined-modality arm. Combined-modality trials employing concurrent chemoradiation have suggested improved loco-regional control resulting in improved survival. These data suggest that both induction and concurrent treatment may be important and may exert their benefit in different manners: induction therapy with effective chemotherapy reduces the rate of overt metastatic disease, while concurrent treatment improves local control by enhancing the local effect of TRT. Four trials to date have been published addressing sequential versus concurrent therapy. In these trials, concurrent treatment yielded improved survival over the sequential approach. The value of either induction or consolidation therapy in addition to concurrent chemotherapy is currently being addressed in randomized Phase III trials.

The study will evaluate the incorporation of ZD1839 with concurrent CP and TCRT to a dose of 74 Gy following 2 cycles of induction CIP. The primary objective will be to define the toxicity profile of this approach. With amendment 2, patients will no longer receive maintenance ZD1839. Given the data generated on LCCC 9603 and 2001, this "hybrid" platform of induction CIP followed by concurrent TCRT (74 Gy) and CP seems appropriate for incorporation of ZD1839 because of the general tolerance of this therapy in good PS, unresectable, Stage III NSCLC subjects. Given that esophagitis is the primary toxicity seen with this approach, stopping rules will be in place for excessive esophageal toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older.
2. Subjects with histologically or cytologically confirmed NSCLC that is considered generally unresectable or inoperable. No prior chemotherapy for NSCLC or thoracic radiotherapy is allowed.
3. Subjects with Stage IIIA or IIIB disease (clinically or surgically staged).
4. Subject with disease designated T3, N0-N1 based on mediastinal invasion or proximity to the carina.

   Subjects with contralateral mediastinal disease (N3) are eligible if all gross disease can be encompassed within the radiation port.
5. Subjects with pleural fluid that is a transudate and is cytologically negative.
6. Subjects with pleural effusions that are seen only on CT scan and are too small to tap.
7. Subjects with measurable or evaluable disease.
8. Subjects with PS of 0 or 1 by the ECOG scale (see Appendix 2).
9. Subjects with laboratory values as follows:

   Absolute granulocyte count: ≥1,500/µL Platelets: ≥100,000/µL Total bilirubin: ≤1.5 x institutional upper normal limit Serum creatinine: <1.6 mg/dL or Creatinine clearance:>40 mL/min

   AST and ALT: ≤2.5 x institutional upper normal limit FEV 1 >800 cc
10. Subjects must be nonpregnant and non-lactating. Subjects of childbearing potential must implement an effective method of contraception during the study. All female subjects, except those who are postmenopausal or surgically sterilized, must have a negative pre-study serum or urine pregnancy test.
11. Subjects must have a life expectancy > 2 months.
12. Subjects must be seen by both a medical oncologist and a radiation oncologist before registration.
13. Subjects must be informed of the investigational nature of the study and must sign an informed consent form.

Exclusion Criteria:

1. Subjects with disease designated T3, N0-N1 based on chest wall invasion, subjects with N3 supraclavicular disease, or subjects with superior sulcus tumors.
2. Subjects with cytologically positive pleural effusions.
3. Subjects who have received prior chemotherapy or radiochemotherapy for lung cancer or prior chest radiotherapy.
4. Subjects who are < 3 weeks since formal exploratory thoracotomy.
5. Subjects with a history of other cancers except in situ carcinoma of the cervix or breast, inactive nonmelanomatous skin cancer, or other cancer, unless the subject has been free of disease for > 5 years.

   Also, exceptions can be made by the PI for a subject with a malignancy for which the prognosis is substantially better than the subject's prognosis for NSCLC.
6. Subjects with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment. Subjects with post-obstructive pneumonia remain eligible.
7. Subjects with dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
8. Pregnant or breast-feeding females or subjects not using adequate methods of birth control.
9. Subjects receiving other investigational therapy or non-approved therapy within 30 days before Day 1 of protocol treatment.
10. Subjects with known hypersensitivity to E coli-derived proteins, pegfilgrastim, or any component of the product will be excluded.
11. Subjects with metastatic disease are excluded.
12. Subjects taking phenytoin, rifampicin, barbiturates, carbamazepine, or St. John's Wort.
13. Any evidence of clinically active ILD (subjects with chronic stable radiographic changes who are asymptomatic need not be excluded).
14. Subjects with evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
15. As judged by the investigator, subjects with any evidence of severe or uncontrolled systemic disease (eg, unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
16. Subjects with known severe hypersensitivity to ZD1839 or any of the excipients of this product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-11; Primary Completion 2006-01 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing toxicity | 60 days
  Toxicity of the combination of induction carboplatin/paclitaxel/irinotecan, followed by concurrent carboplatin/paclitaxel/ZD1839 and high-dose TCRT, will be assessed by CTCAE criteria
Efficacy of 2 cycles of induction paclitaxel/carboplatin/irinotecan | 42 days
  To estimate the efficacy of 2 cycles (42 days) of induction paclitaxel/carboplatin/irinotecan, followed by concurrent carboplatin/paclitaxel/ZD1839 using RECIST criteria to evualate tumor response.

SECONDARY OUTCOMES:
Progression Free Survival | 5 years
  Radigraphic response measured by RECIST critera.

CONTACTS AND LOCATIONS:
Overall Officials: David Morris, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States